CLINICAL TRIAL: NCT05460936
Title: Effects of Lower Extremity Functional Training (LIFT) on Gross Motor Function and Gait in Children With Spastic Cerebral Palsy
Brief Title: Lower Extremity Functional Training (LIFT) on Gross Motor Function and Gait in Children With Spastic CP
Acronym: LIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR& AHS /22/0715
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy. gait training, motor learning, functional training, balance, hemiplegic gait.
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physical therapy (Active Comparator): Resistive Exercises Stretching exercise of quadriceps , hamstring adductors and abductors.
  Interventions: Other: conventional physical therapy
- Lower Extremity Functional Training (Experimental): motor learning, skill progression, and resistance training to target the balance, strength, and coordination impairments of the lower extremities. Motor learning will be based on strength and balance training using tandem walks, balance boards, and one-leg standing. Skill progression will be used to challenge the LIFT and the strength training will be achieved by performing sit-to-stand, sit-ups, stair climbs, and vertical jumps
  Interventions: Other: Lower Extremity Functional Training

INTERVENTIONS:
Other: Lower Extremity Functional Training — motor learning, skill progression, and resistance training to target the balance, strength, and coordination impairments of the lower extremities. Motor learning will be based on strength and balance training using tandem walks, balance boards, and one-leg standing. Skill progression will be used to challenge the LIFT and the strength training will be achieved by performing sit-to-stand, sit-ups, stair climbs, and vertical jumps
  Arms: Lower Extremity Functional Training
Other: conventional physical therapy — Resistive Exercises Stretching exercise of quadriceps , hamstring adductors and abductors.
  Arms: conventional physical therapy

SUMMARY:
Cerebral Palsy is a developmental disorder caused by damage to the brain before, during or after birth. Spastic Cerebral Palsy is one of the most common types of cerebral Palsy. It affects about 80% of cerebral palsy. Spastic CP is characterized by increased muscle tone, jerky movements, joint stiffness, and muscle tightness. Spastic Cerebral primarily affects strength, coordination, and balance resulting in gait difficulties and affecting gross motor functioning. These abnormalities affect the very basic activities of daily life (ADLs). Even if the child is able to walk the motor skills are usually disturbed which are very important to improve and maintain gross motor functioning. Physical therapy plays a vital role in overcoming these issues.

DETAILED DESCRIPTION:
In the previous studies the effects of LIFT on the trunk and core has been studies however, the data on the effects on the gross motor skills are very less. In addition to that the effects of lower extremity functional training on the gait have also been limited to a few studies only. The past studies were of very short time period due to which the proper effects of LIFT on the gait and gross motor skills were not very well understood.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not able to stand
* Age between 7 to 16 years
* Patients living near the designated center

Exclusion Criteria:

* Patients with comorbidities
* Patients with cognitive impairment
* Patients who are not able to follow commands
* Patients with a history of falls

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
1-minute walk test | 8th week
  1-minute walk test will be used to measure the functional ability of the child. This is a cost-effective and user-friendly tool which makes it a very suitable tool to be used in various clinical settings. This tool is selected because of the low attention span and ability of children to perform other tests. This test can be conducted in a short duration of time giving the required results
Single leg stance | 8th week
  a. The single-leg stance test is used to check the balance control along with the static posture control on the affected side. This tool is considered valuable and effective in monitoring the musculoskeletal; status and neurological status of the individual
Gross Motor Function Measurement | 8th Week
  The Gross Motor Function Measure31 is a criterion-referenced assessment designed to be used with children with cerebral palsy. It evaluates the child's ability to complete motor functions, such as rolling, crawling, sitting, standing, walking, running, stair use, and jumping.

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, PhD, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - International Therapy Services Center, Lahore, Punjab Province
  - Rising Sun Institute, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baldon Rde M, Serrao FV, Scattone Silva R, Piva SR. Effects of functional stabilization training on pain, function, and lower extremity biomechanics in women with patellofemoral pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):240-251, A1-A8. doi: 10.2519/jospt.2014.4940. Epub 2014 Feb 25. PMID 24568258
- [Background] Vereijken A, Aerts I, Jetten J, Tassignon B, Verschueren J, Meeusen R, van Trijffel E. Association between Functional Performance and Return to Performance in High-Impact Sports after Lower Extremity Injury: A Systematic Review. J Sports Sci Med. 2020 Aug 13;19(3):564-576. eCollection 2020 Sep. PMID 32874110
- [Background] Bowman EN, Elshaar R, Milligan H, Jue G, Mohr K, Brown P, Watanabe DM, Limpisvasti O. Proximal, Distal, and Contralateral Effects of Blood Flow Restriction Training on the Lower Extremities: A Randomized Controlled Trial. Sports Health. 2019 Mar/Apr;11(2):149-156. doi: 10.1177/1941738118821929. Epub 2019 Jan 14. PMID 30638439